CLINICAL TRIAL: NCT03282565
Title: Functional Resistance Training During Gait: A Novel Intervention to Improve Knee Knee Function After ACL Reconstruction
Brief Title: Functional Resistance Training to Improve Knee Function After ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Riann Palmieri-Smith, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00133860; R21HD092614 (NIH)
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Results first posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: ACL; Quadriceps; Muscle; Resistance Training
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Braces

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Functional Resistance Training with a Brace (Experimental): Participants will receive functional resistance training via a knee brace while walking on a treadmill 2-3 times a week for about 8 weeks.
  Interventions: Other: Functional Resistance Training with Brace
- Functional Resistance Training with Elastic Band (Experimental): Participants will receive functional resistance training via an elastic band attached at the ankle while walking on a treadmill 2-3 times a week for about 8 weeks.
  Interventions: Other: Functional Resistance Training with Elastic Band
- Control (Sham Comparator): Participants will while on a treadmill without an applied resistance 2-3 times a week for about 8 weeks.
  Interventions: Other: Control

INTERVENTIONS:
Other: Functional Resistance Training with Brace — A brace will be strapped to the leg and apply resistance across the knee while subjects walk on a treadmill.
  Arms: Functional Resistance Training with a Brace
Other: Control — A brace will be strapped to the leg and will not apply resistance across the knee while subjects walk on a treadmill.
  Arms: Control
Other: Functional Resistance Training with Elastic Band — An elastic band will be strapped to the leg and apply resistance across the knee while subjects walk on a treadmill.
  Arms: Functional Resistance Training with Elastic Band

SUMMARY:
The purpose of this study is to examine if thigh muscle weakness and the lack of muscle activation that accompanies ACL injury and reconstruction can be improved with functional resistance training.

DETAILED DESCRIPTION:
Profound quadriceps weakness is ubiquitous after anterior cruciate ligament (ACL) reconstruction, and current rehabilitation approaches are not successful in optimizing quadriceps strength and knee function even years after the surgery. We hypothesize that suboptimal strength and functional outcomes after ACL surgery are due to the lack of task-specific exercise elements during strength training. This application seeks to assess whether progressive functional resistance training during gait will significantly improve quadriceps function, neural excitability, and knee mechanics during gait. The proposed studies will not only lay the foundation for a novel training paradigm, but will also improve our understanding of the mechanisms mediating neuromuscular and biomechanical changes after functional resistance training.

ELIGIBILITY:
Inclusion Criteria:

* aged 14-40 years
* suffered an acute, complete ACL rupture
* willingness to participate in testing and follow-up as outlined in the protocol
* English-speaking

Exclusion Criteria:

* inability to provide written informed consent
* female subjects who are pregnant or are planning to become pregnant
* previous ACL injury
* previous surgery to either knee
* bony fracture accompanying ACL injury
* patients who experienced a knee dislocation;
* patients who are contraindicated for transcranial magnetic stimulation (e.g., metal implants in head, unexplained recurrent headaches, history of seizures, epileptogenic drugs, active psychiatric illness, etc.).

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-17 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Riann Palmieri-Smith, PhD, Principal Investigator — University of Michigan; Chandramouli Krishnan, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Functional Resistance Training With Brace: Participants received functional resistance training while walking on a treadmill 2-3 times a week for 8 weeks.
  Functional Resistance Training: A customized knee brace was strapped to the leg and applied resistance during knee flexion and extension while subjects walked on a treadmill.
- Functional Resistance Training With Elastic Band: Participants received functional resistance training while walking on a treadmill 2-3 times a week for 8 weeks.
  Functional Resistance Training: An elastic band strapped to the ankle provided resistance during knee extension while subjects walked on a treadmill.
- Control: Participants walked on a treadmill without an applied resistance 2-3 times a week for about 8 weeks.
  Control: A knee brace was strapped to the leg and did not apply resistance while subjects walked on a treadmill.
Period: Overall Study
Arm/Group | Functional Resistance Training With Brace | Functional Resistance Training With Elastic Band | Control
Started | 10 | 10 | 10
Completed | 10 | 8 | 8
Not Completed | 0 | 2 | 2
Not completed — COVID-19 Research Shutdown | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Functional Resistance Training With Brace | Functional Resistance Training With Elastic Band | Control | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.8 (6.2) | 22.1 (4.5) | 20.4 (5.6) | 20.4 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 18
  Male | 4 | 4 | 4 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 3
  White | 9 | 7 | 8 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30
Height [Mean (Standard Deviation); unit: centimeters] | 174 (11.2) | 172.3 (7.9) | 169.8 (9.0) | 172.0 (9.4)
Mass [Mean (Standard Deviation); unit: kilograms] | 70.1 (10.5) | 70.3 (12.2) | 70.2 (13.3) | 70.2 (12.0)
Time Since Surgery to Baseline Study Testing [Mean (Standard Deviation); unit: weeks] | 8.9 (2.6) | 9.5 (2.5) | 10.3 (3.1) | 9.6 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Quadriceps Muscle Strength
Description: Isometric quadriceps strength was measured with the knee at 60 degrees using an isokinetic dynamometer prior to the intervention and immediately after the intervention. Post-test minus pre-test change scores were calculated.
Time Frame: Pre-test measurements were taken at ~9-10 weeks after ACL reconstruction and Post-test measurements were taken at ~18-20 weeks after ACL reconstruction.
Measure: Mean (Standard Error); unit: Nm/Kg
Arm/Group | Functional Resistance Training With Brace | Functional Resistance Training With Elastic Band | Control
Number analyzed (Participants) | 10 | 9 | 9
Nm/Kg | .674 (.124) | .398 (.130) | .279 (.130)

2. Secondary Outcome: Quadriceps Voluntary Activation
Description: Quadriceps voluntary activation was measured using the burst superimposition technique and calculated using the central activation ratio (CAR). The CAR formula is calculated using the peak torque generated immediately prior to the delivery of the stimulus (or the maximum voluntary isometric contraction, MVIC) being divided by the peak torque generated as a result of the electrical stimulus (MVIC plus superimposed burst) and then multiplied by 100. Equation is: MVIC/(MVIC + superimposed burst) × 100. A CAR of 100 represents complete volitional quadriceps activation.
  Voluntary activation was quantified immediately after the intervenapproximately 9-10 weeks after the int from baseline to the end of intervention will be assessed and compared between groups.
Time Frame: Immediately after the intervention or approximately 18-20 weeks after ACL reconstruction
Measure: Mean (Standard Error); unit: percentage of activation
Arm/Group | Functional Resistance Training With Brace | Functional Resistance Training With Elastic Band | Control
Number analyzed (Participants) | 10 | 9 | 9
percentage of activation | 73.19 (6.56) | 69.55 (7.72) | 68.29 (7.19)

3. Secondary Outcome: Knee Flexion Angle Symmetry
Description: The knee flexion angle (measured in degrees) during the stance phase was gathered for both limbs using three dimension motion capture and recorded while subjects walked overground. A knee flexion angle symmetry score was computed using the following formula: ensemble average of knee flexion angle of ACL limb minus the ensemble average of knee flexion angle of the non-ACL limb. The mean difference between pre-intervention and post-intervention (post minus pre) knee flexion symmetry scores were calculated for each group. Higher values suggest greater increases in knee flexion angle symmetry from pre-intervention to post-intervention.
Time Frame: Pre-intervention values were recorded at ~9-10 weeks after ACL reconstruction and before the start of the intervention. Post-intervention values were recorded after the 8-week intervention (~18-20 weeks after ACL reconstruction)
Measure: Mean (95% Confidence Interval); unit: Angle Symmetry (degrees)
Arm/Group | Functional Resistance Training With Brace | Functional Resistance Training With Elastic Band | Control
Number analyzed (Participants) | 9 | 8 | 9
Angle Symmetry (degrees) | 3.230 [0.658 to 5.803] | 0.556 [-0.857 to 1.970] | 0.846 [-0.917 to 2.608]

4. Secondary Outcome: Knee Moment Symmetry
Description: The sagittal plane knee moment (units Nm) during the stance phase was gathered for both limbs using three dimensional motion capture and recorded while subjects walk overground. A symmetry score was computed using the following formula: ensemble average of the knee moment of the ACL limb (Nm) - ensemble average of the knee moment of the non-ACL limb (Nm). The mean difference between pre-intervention and post-intervention knee moment symmetry scores (post minus pre) were calculated for each group. Higher values represent the greater increases in knee moment symmetry from pre-intervention to post-intervention.
Time Frame: Pre-intervention scores were recorded prior to the start of the intervention and approximately 9-10 weeks after ACL reconstruction. Post-intervention scores were recorded after the 8 week intervention or approximately 18-20 weeks after ACL reconstruction
Measure: Mean (95% Confidence Interval); unit: Moment Symmetry (Nm)
Arm/Group | Functional Resistance Training With Brace | Functional Resistance Training With Elastic Band | Control
Number analyzed (Participants) | 9 | 8 | 9
Moment Symmetry (Nm) | .0144 [-0.057 to 0.086] | 0.132 [0.0408 to 0.224] | -0.042 [-0.078 to -0.0074]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the course of the study. The timeframe of the study was approximately 5 months. Adverse events during a period from about 8 weeks after ACL reconstruction to about 28 weeks after reconstruction.
Description: Does not differ from clinical trials.gov
Arm/Group | Functional Resistance Training With Brace | Functional Resistance Training With Elastic Band | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT03282565/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT03282565/ICF_001.pdf